CLINICAL TRIAL: NCT00440362
Title: A Single-Site, Phase 1/2, Double-Blind, Safety and Immunogenicity Trial of an Alphavirus Replicon Vaccine Expressing Influenza A/Wyoming/03/2003 Hemagglutinin (AVX502) in Healthy Volunteers
Brief Title: A Phase 1/2 Clinical Trial of an Alphavirus Replicon Vaccine for Influenza
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AlphaVax, Inc. (Industry)
Responsible Party: Robert Olmsted, Ph.D., AlphaVax, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AVX502-002
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Last update posted 2008-11-10 (Estimated); Status verified 2008-11

CONDITIONS: Influenza
Keywords: Influenza; Flu; A/Wyoming/03/2003; Alphavirus
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- T1 (Active Comparator)
  Interventions: Biological: AVX502
- T2 (Active Comparator)
  Interventions: Biological: AVX502
- T3 (Active Comparator)
  Interventions: Biological: AVX502
- T4 (Active Comparator)
  Interventions: Biological: AVX502
- T5 (Active Comparator)
  Interventions: Biological: AVX502
- T6 (Active Comparator)
  Interventions: Biological: AVX502
- T7 (Active Comparator)
  Interventions: Biological: AVX502
- T8 (Active Comparator)
  Interventions: Biological: AVX502
- C1 (Placebo Comparator)
  Interventions: Biological: Placebo
- C2 (Placebo Comparator)
  Interventions: Biological: Placebo
- C3 (Placebo Comparator)
  Interventions: Biological: Placebo
- C4 (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AVX502 — 1 dose at 2e8 IU given at t=0 via IM route
  Arms: T2
Biological: AVX502 — 1 dose at 2e7 IU given at T=0 via the IM route
  Arms: T1
Biological: AVX502 — 1 dose at 2e7 IU given at t=0 via the SC route
  Arms: T3
Biological: AVX502 — 1 dose at 2e8 IU given at T=0 via the SC route
  Arms: T4
Biological: AVX502 — 2 doses at 2e7 IU given at T=0 and 8 weeks via the IM route
  Arms: T5
Biological: AVX502 — 2 doses at 2e8 IU given at T=0 and 8 weeks via the IM route
  Arms: T6
Biological: AVX502 — 2 doses of 2e7 IU given at t=0 and 8 weeks via the SC route
  Arms: T7
Biological: AVX502 — 2 doses at 2e8 IU given at T=0 and 8 weeks via the SC route
  Arms: T8
Biological: Placebo — 1 dose of placebo given at T=0 via the IM route
  Arms: C1
Biological: Placebo — 1 dose of placebo given at T=0 via the SC route
  Arms: C2
Biological: Placebo — 2 doses of placebo given at T=0 and 8 weeks via the IM route
  Arms: C3
Biological: Placebo — 2 doses of placebo given at T=0 and 8 weeks via the SC route
  Arms: C4

SUMMARY:
AVX502, an alphavirus replicon vaccine expressing an influenza HA protein, is a candidate vaccine against influenza.

The objectives of this Phase 1 study are to test the safety of the vaccine and the immune response to the vaccine in healthy volunteers 18-40 years of age. Volunteers will be assigned by randomization to receive either the vaccine or an inactive substance (placebo) by injections in each arm on one or two occasions over 2 months. The study will last 4 months and will have a total of 8 visits.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase 1/2 study of the safety and immunogenicity of AVX502 vaccine at two dosage levels and two routes of administration in healthy volunteers conducted at a single research center. A total of 216 participants will be enrolled. Participants will be randomized to receive active vaccine at one of two dosage levels or placebo in a 4:4:1 ratio. Within each active dosage level or placebo subgroup, participants will be randomized to receive their injections by either IM or SC injection in a 1:1 ratio, and will also be randomized to receive either 1 injection (at Week 0) or 2 injections (1 at each of two visits at Weeks 0 and 8) in a 1:1 ratio. Vaccine will be administered by a study nurse in an outpatient setting and all participants will be followed for 4 months after the first immunization. Safety data will include local and systemic reactogenicity after each dose of vaccine, collected in a systematic format using a subject memory aid and a standard grading scale, specific safety laboratory parameters and general AEs. Immunogenicity data will be obtained by collecting blood at defined time points before and after immunization and separating serum (for measurement of antibodies to HA by ELISA and hemagglutination inhibition assays and to the vaccine vector by a VRP neutralization assay) and peripheral blood mononuclear cells (PMBC) (for measurement of cellular immune responses to HA peptides).

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 40 years of age, inclusive;
2. Good general health without significant physical examination findings or clinically significant abnormal laboratory results;
3. Available to participate for the entire study period of approximately 4 months;
4. For women of childbearing potential, a negative urine pregnancy test at screening and before each immunization, and agreement to consistently use contraception from 28 days prior to enrollment until the last protocol visit, for sexual activity that could lead to pregnancy;
5. Acceptable laboratory parameters: hemoglobin ≥ 11.2 g/dL for women, ≥ 12.8 g/dL for men, white blood cell count 3,300 - 12,000 cells/mm3, platelet count 125,000 - 550,000/mm3, alanine aminotransferase (ALT) within normal range for study laboratory, serum creatinine within normal range for study laboratory, normal urine dipstick (negative glucose, negative hemoglobin, and negative or trace protein), negative hepatitis B virus (HBV) and hepatitis C virus (HCV) blood tests, negative HIV blood test;
6. Willingness to have blood stored for up to 10 years for use in additional assays to evaluate immune responses to influenza or the alphavirus vector if such assays become available
7. Willingness to participate in the study as evidenced by signed informed consent obtained before screening.

Exclusion Criteria:

1. Venous access deemed inadequate for the phlebotomy demands of the study;
2. Women who are breast feeding;
3. In female subjects, a positive urine pregnancy test at screening or on the day of any vaccine injection;
4. Receipt of any influenza vaccine within 12 months prior to enrollment;
5. Receipt of any other vaccine within 30 days prior to enrollment;
6. Use of any investigational agent within 30 days prior to enrollment;
7. Receipt of immunoglobulin or blood products within 60 days prior to enrollment;
8. Use of cytotoxic medications within 6 months prior to enrollment;
9. Use of systemic corticosteroids within 6 months prior to enrollment (except that participants who have completed a course of prednisone, at up to 20 mg per day for up to 7 days, at least 1 month prior to enrollment are eligible for enrollment);
10. Presence of any factor that places the individual at increased risk for severe complications from influenza;
11. History of serious adverse reactions to any vaccine, including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema or abdominal pain;
12. History of autoimmune disease;
13. History of splenectomy;
14. History of malignancy within the last 3 years (except that participants with a diagnosis of basal cell carcinoma of the skin are eligible for enrollment);
15. Psychiatric condition that may interfere with the ability to comply with the protocol requirements. Specifically excluded are persons with history of psychosis within the past 3 years or history of suicidal attempt or gesture within the past 3 years;
16. History of medical, occupational or family problems as a result of alcohol or illicit drug use during the past 12 months;
17. Any condition which leads the investigator to believe that the participant cannot comply with the protocol requirements or that may place the participant at an unacceptable risk for participation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2007-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Evaluate safety of AVX502 in healthy volunteers via frequency of Grade 2-4 systemic reactogenicity events, grade 3 or 4 local vaccine reactions and all AE's | 16 weeks

SECONDARY OUTCOMES:
Evaluate immunogenicity of AVX502 in healthy volunteers via serum antibody concentration | 4 weeks post first dose of vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Olmsted, Ph.D., Principal Investigator — AlphaVax, Inc.
Locations (1):
- Johnson County Clin-Trials, Lenexa, Kansas, United States

REFERENCES:
- See also: AlphaVax, Inc. — http://www.alphavax.com
- See also: Johnson County Clin-Trials — http://www.jococt.com